CLINICAL TRIAL: NCT07154563
Title: Rapid Assessment of Sentinel Lymph Node Metastasis Status Using a Pan-CK-targeting NIR-II Fluorescent Probe in Breast Cancer
Acronym: NIR-II
Status: Recruiting | Type: Observational
Sponsor: Yunnan Cancer Hospital (Other)
Collaborators: Xiang'an Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLX2025-060
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Metastatic; Sentinel Lymph Node; Sentinel Lymph Node Biopsy (SLNB); Metastasis
Keywords: NIR-II; Breast Cancer; Sentinel Lymph Node; Metastasis
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NIR-II probe incubation: NIR-II probe incubation Group/Cohort Description: Freshly excised SLNs will be fully immersed in NIR-II probe ((i.e:ICG-CK) incubation solution (6.25, 12.5, 25, 50, 100 ug/mL) for 1, 3, 5, 7, or 10 min, then rinsed with PBST buffer for 5 min and dried with absorbent paper. NIR-II fluorescence imaging will then be performed under the DPM NIR-II system. The correlation between pathological features and fluorescence information will be further analyzed.
  Interventions: Diagnostic Test: NIR-II probe (i.e ICG-CK) incubation solution

INTERVENTIONS:
Diagnostic Test: NIR-II probe (i.e ICG-CK) incubation solution — After incubating the lymph node tissue with an optimal concentration of NIR-II probe for an appropriate amount of time, the tissue is washed with eluent, and then the fluorescence intensity of different tissues is detected to assess whether the tissue has cancer tissue invasion.

SUMMARY:
Breast malignant tumors are a serious threat to women's health, and the current treatment for breast malignant tumors is still dominated by surgery, but the problems faced by patients after surgery such as edema and tumor recurrence are still relatively common, and the high recurrence rate and the occurrence of postoperative complications are closely related to the removal of metastatic lymph nodes during surgery. Therefore, accurate assessment of sentinel lymph node (SLN) metastases is essential to determine the extent of axillary lymph node dissection (ALND) and minimize complications. In this study, we developed a new technique that can rapidly distinguish between metastatic lymph nodes and normal sentinel lymph nodes (SLNs) in breast cancer patients. Briefly, fresh tissue is incubated with the probe and imaged immediately after intraoperative sentinel lymph node resection to identify the metastatic status of SLN. The accuracy of fluorescence imaging is confirmed by pathological diagnosis.

DETAILED DESCRIPTION:
Following patient enrollment, surgical interventions were performed in accordance with standardized clinical protocols. During the operative procedure, the excised sentinel lymph nodes (SLNs) underwent specialized incubation processing. The detailed experimental protocol was conducted as follows:

1. Preparation of incubation solution The molecular probe was reconstituted in phosphate-buffered saline (PBS) to create incubation solutions with concentration gradients of 6.25, 12.5, 25, and 50 μg/mL. Solution preparation was performed at ambient temperature under light-protected conditions.
2. Ex vivo SLN tissue incubation Freshly excised SLN specimens were fully immersed in the prepared solutions for designated durations (1, 3, 5, 7, or 10 minutes). Subsequent processing included a 5-minute wash cycle with PBST buffer (0.05% Tween 20 in PBS) followed by blot-drying using absorbent filter paper.
3. NIR-II fluorescence imaging analysis Imaging acquisition was conducted using the Digital Precision Medicine (DPM) NIR-II system. Following initial system parameter calibration and spatial scaling, fluorescence signals were captured and quantitatively analyzed to determine SLN metastatic status through proprietary diagnostic algorithms.
4. Histopathological validation Final diagnostic confirmation was obtained through comprehensive histopathological examination conducted by certified pathologists.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18-75 years of age
* Patients presenting with a breast nodule or mass presumed to be resectable on pre-operative assessment
* Breast cancer patients who are scheduled to undergo sentinel lymph node biopsy or axillary lymph node dissection;
* Good operative candidate
* Subject capable of giving informed consent and participating in the process of consent

Exclusion Criteria:

* Patients unable to participate in the consent process
* Patients had contraindications to surgery, such as serious cardiopulmonary disease, coagulation dysfunction, etc

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to enroll 90 female patients, aged 18 to 75 years, who have been assessed to have resectable breast nodules or masses and are scheduled to undergo surgery. During the surgery, the resected lymph nodes will be incubated with theNIR-II probe(ICG-CK) solution, and NIR-II fluorescence signals from the tissues will be collected.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Uptake of the dye by the tissue(i.e metastatic SLN) | 1 year
  Ability of the imaging system to discern the uptake of the dye by the metastatic SLN . Detected with imaging probe.
False positive rates of the NIR-II probe (ICG-CK) | 1 year
  Microscopic examination and immunohistochemistry of tumor performed by a pathologist. This will allow investigators to compare pathology results with fluorescence images taken by imaging probe to calculate false positive (i.e., identification of non metastatic SLN) rates of ICG-CK.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan 650118, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39413161/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37540231/